CLINICAL TRIAL: NCT00158288
Title: LAAM With Behavioral Treatment for Opioid/Cocaine Abuse
Brief Title: The Efficacy of Methadyl Acetate (LAAM) and Contingency Management Procedures for Treating Dual Opioid and Cocaine Abuse - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Yale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09876-1; R01-09876-1
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2005-09

CONDITIONS: Behavior Therapy; Cocaine; Contingency Management; Heroin Dependence; LAAM; Opioid Dependence; Substance-Related Disorders; Alcohol & Drug Use
Keywords: Substance Use Disorders
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders; Substance-Related Disorders | interventions — Methadyl Acetate

INTERVENTIONS:
Behavioral: LAAM

SUMMARY:
Although LAAM, a derivative of methadone, has been successfully used as an alternative to methadone maintenance in opioid addicts, its effect on concurrent opioid and cocaine abuse has not been ascertained. Thus, this study proposes to examine the clinical efficacy of low- and high-dose LAAM maintenance on opioid and cocaine use in opioid-dependent cocaine abusers. In addition, since contingency management procedures have demonstrated some success in decreasing cocaine use in cocaine-abusing individuals, this study also proposes to examine the clinical efficacy of the presence or absence of contingency management procedures targeting illicit drug use.

DETAILED DESCRIPTION:
One hundred forty male and female opioid-dependent cocaine abusers will be stratified by sex and randomly assigned to one of four treatment groups according to a 2 x 2 experimental design: low-dose LAAM (99 mg/wk) with adjunct contingency management procedures; low-dose LAAM (99 mg/wk) without adjunct contingency management procedures; high-dose LAAM (330 mg/wk) with adjunct contingency management procedures; and high-dose LAAM (330 mg/wk) without adjunct contingency management procedures. The duration of the study will be 24 weeks, with LAAM being administered on a thrice-weekly (MWF) basis.

Subjects are inducted onto LAAM during weeks 1-3 and then maintained on their assigned maintenance dose (99 mg/wk or 330 mg/wk) through week 24. During maintenance, the Friday dose will be 1.3 times greater than the Monday and Wednesday dose. At the conclusion of the study, subjects undergo detoxification from LAAM over a 4-week period. For those in the contingency management procedure group, each drug-free urine submitted will result in a voucher worth a certain monetary value that increases for consecutively drug-free urines (weeks 1-12) or a monetary voucher with a fixed value (weeks 13-24). Subjects not assigned to the contingency management procedure will receive monetary vouchers (weeks 1-24) according to a yoked-control schedule (that is, not contingent upon illicit drug abstinence). Vouchers can be exchanged for mutually agreed upon goods and services at any time during the study. Outcome measures will include: 1) treatment retention, 2) illicit drug use, 3) self-reported adverse and opioid withdrawal symptoms, and 4) psychosocial functioning. Follow-up interviews at nine months and/or one year post-study entry will be conducted to determine status post-treatment. Prognostic factors (i.e., sex, post-traumatic stress disorder, and depression), will also be examined in relation to treatment outcome and post-treatment status.

ELIGIBILITY:
Inclusion Criteria:

* One hundred forty male and female cocaine-abusing, opioid-dependent individuals between the ages 21-55, with at least 40% women and 40% Afro-Americans, who not be currently enrolled in treatment, will be entered into the study. Subjects must have current opioid dependence as evidenced by documentation of prior treatment for opioid dependence or signs of withdrawal upon administration of naloxone (0.8 mg, i.m.), and opioid-positive urine screen. Subjects also must be current users of cocaine with self-reported use of > 12 gms during the preceding 12 months, self-reported use of > 1 gm/week in the month preceding study entry, and cocaine-positive urine screen. Subjects must fulfill DSM-III-R criteria for opioid and cocaine dependence. These criteria will be ascertained using the substance abuse section of the SCID interview developed for use with DSM-III-R

Exclusion Criteria:

* Criteria for exclusion include current diagnosis of other drug or alcohol dependence (other than opiates, cocaine or tobacco); ill health (e.g., major cardiovascular, renal, endocrine, hepatic disorder); respiratory condition (e.g., asthma); history of major psychiatric disorder (psychosis, schizophrenia, bipolar, major depression); current suicidality; LFT's (i.e., liver enzymes) greater than 3 times normal levels; and pregnancy.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140
Dates: Start 1997-03; Study Completion 2001-08

PRIMARY OUTCOMES:
Urine toxicology for cocaine

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, Ph.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Result] Oliveto A, Poling J, Sevarino KA, Gonsai KR, McCance-Katz EF, Stine SM, Kosten TR. Efficacy of dose and contingency management procedures in LAAM-maintained cocaine-dependent patients. Drug Alcohol Depend. 2005 Aug 1;79(2):157-65. doi: 10.1016/j.drugalcdep.2005.01.007. PMID 16002025